CLINICAL TRIAL: NCT04642222
Title: APOLO-Teens, a Web-based Intervention For Treatment-seeking Adolescents With Overweight/Obesity: A Multicenter Randomized Controlled Trial
Brief Title: APOLO-Teens, a Web-based Intervention For Adolescents With Overweight/Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Eva Conceição, Research Fellow, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SECVS 142/2015; POCI-01- 0145-FEDER-028209 (Other Grant/Funding Number: Fundação Para a Ciência e Tecnologia)
Record Dates: First submitted 2020-11-17; First posted 2020-11-24 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Pediatric Obesity
Keywords: Adolescent; Web-based intervention; Health promotion; Eating Behaviors
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a randomized control trial with two groups: the Treatment As Usual control group (TAU group) and the APOLO-Teens web-based intervention group (APOLO-Teens group). Adolescents attending a medical appointment scheduled for any multidisciplinary obesity appointment at a public Portuguese health facility will be invited to participate. The criteria for inclusion/exclusion will be given to the healthcare professionals conducting these medical appointments, to screen for potential participants. After completing the baseline assessment participants will be consecutively randomized to the Treatment As Usual control group (TAU group) or the APOLO-Teens web-based intervention group (APOLO-Teens group). Participants in the APOLO-Teens group received the APOLO-Teens web-based intervention in addition to their treatment as usual (TAU).
Who Masked: Outcomes Assessor
Masking Description: Randomization is performed by a researcher not involved in data management. The researcher who evaluates the outcomes of interest is masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APOLO-Teens Intervention Group (APOLO-Teens group) (Experimental): In addition to the Treatment As Usual for pediatric obesity offered in Portuguese public hospitals, participants in this group receive the APOLO-Teens web-based intervention. It comprises three key components: 1) a manualized psychoeducational intervention implemented via Facebook® private groups, including cognitive-behavioral therapy strategies; 2) A weekly self-monitoring system (the APOLO-Teens web application) with automatic feedback messages assessing hours of physical activity, sedentary time, and consumption of fruits and vegetables; and 3) Monthly chat sessions.
  Interventions: Behavioral: APOLO-Teens web-based intervention
- Treatment As Usual (TAU) Control Group (TAU control group) (Active Comparator): Treatment As Usual control group receives the standard intervention for pediatric obesity offered in Portuguese public hospitals. It comprises pediatric or/and nutritional appointments, usually a 30-minute appointment every 3 months. These appointments usually include a physical examination (weight, height) and personalized dietary/lifestyle recommendations. The Treatment As Usual intervention is common to the APOLO-Teens group and TAU control groups.
  Interventions: Other: Treatment as Usual for Pediatric Obesity

INTERVENTIONS:
Behavioral: APOLO-Teens web-based intervention — The APOLO-Teens web-based intervention is a 6-month cognitive-behavioral lifestyle program developed to optimize treatment as usual for pediatric obesity in public portuguese hospitals.
  Arms: APOLO-Teens Intervention Group (APOLO-Teens group)
Other: Treatment as Usual for Pediatric Obesity — Treatment as Usual for pediatric obesity in portuguese public hospitals.
  Arms: Treatment As Usual (TAU) Control Group (TAU control group)

SUMMARY:
With the demand for weight-loss interventions likely to continue its upward trend over the next decades, the question remains on how to continuously monitor and support overweight and obese adolescents, particularly in the long-term. Moreover, as the burden of the obesity rates increases in health care centers, the development of alternative delivering strategies gains attention. In an environment of limited resources, the development of new-technology based programs seems a promising area to deliver cost-effective interventions to a wide number of individuals. However, the existing studies present several limitations and a challenging aspect of treating obesity in adolescents is the presence of high rates of disordered eating behaviors.

The objective of this study is to develop and test the effectiveness of a web-based Cognitive Behavioral Therapy intervention, for adolescents with overweight/obesity. A Randomized Controlled Trial will compare a control group receiving medical treatment as usual (TAU), and an intervention group receiving TAU plus a psychological/behavioral intervention delivered via the internet.

DETAILED DESCRIPTION:
This research project intends to examine the effectiveness of a Cognitive Behavioral Therapy and psychoeducational based program for adolescents with overweight and obesity delivered as a web-based intervention: APOLO-Teens. Therefore, a randomized controlled trial will compare a control group receiving medical treatment as usual for pediatric obesity in public health care centers in Portugal, and an intervention group receiving TAU plus the APOLO-Teens web-based intervention.

The APOLO-Teens web-based intervention was designed to optimize treatment as usual for pediatric obesity, promoting the adoption of healthy eating habits and lifestyle behaviors. Particularly it aims to promote higher consumption of fruits and vegetables, increase physical activity levels, reduce sedentary time, enhance psychological well-being, and facilitating weight loss.

All participants will be assessed at baseline, 3 months after the beginning of the research protocol/intervention, end of the web-based intervention, and at 6 and 12 months follow-up. All the assessments will be conducted in Qualtrics: Online Survey Software. Repeated Paired Samples T-test will explore differences between the two groups across the assessment times. Multiple linear regression analysis will be applied to explore predictors of weight loss and weight regain, and survival analyses to identify participants with the highest probability to regain weight. Additionally, 3-Level Hierarchical Linear Models will be conducted to explore the temporal occurrence and patterns of change of eating-related variables, physical activity, and BMI z-score in participants from the two groups.

It is expected that the intervention group participants will present a higher frequency of healthy food consumption (fruit/vegetables) and increased physical activity levels at the end of the web-based intervention when compared with TAU group participants. We further expect, differences between the groups regarding eating behavior-related variables, as well as in the psychological features assessed throughout the different assessment points, and ultimately in weight maintenance or regain, with the intervention group presenting lower scores/weight.

ELIGIBILITY:
Inclusion Criteria:

* Participants with overweight or obesity (BMI z-score ≥ 1/BMI percentile ≥ 85th);
* Enrolled in ambulatory treatment for overweight/obesity in a public Portuguese health care center;
* Having a Facebook® account;
* Having access to the Internet at least three times per week.

Exclusion Criteria:

* Medical conditions that affect weight;
* Intellectual disabilities (Specific learning difficulties that prevented adolescents from reading and understanding written text);
* Ambulatory movement limitations (e.g., use of the walking stick, morpho-functional alterations as lower limb amputation, etc.);
* Not being under other interventions for weight loss at the time of enrollment.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Foods/beverages intake | Change from baseline, to 3 months after the begging if the intervention, end of intervention (after 6-months of baseline assessment), 6 and 12 months follow-up. Specific duration of time over which participant change is assessed: 18 months.
  Food/beverages frequency questionnaire, which assesses the frequency of soup, fruit, vegetables on the plate, sweetened beverages drinks and pastries/sweets intake in the previous week.
Minutes of moderate-to-vigorous physical activity per week at school | Change from baseline, to 3 months after the begging if the intervention, end of intervention (after 6-months of baseline assessment), 6 and 12 months follow-up. Specific duration of time over which participant change is assessed: 18 months.
  Youth Activity Profile (YAP): This is a 15 items questionnaire to evaluate psychical activity and sedentary behaviors in youth on the previous seven days.
Minutes per week spent in sedentary behaviors | Change from baseline, to 3 months after the begging if the intervention, end of intervention (after 6-months of baseline assessment), 6 and 12 months follow-up. Specific duration of time over which participant change is assessed: 18 months.
  Youth Activity Profile (YAP): This is a 15 items questionnaire to evaluate psychical activity and sedentary behaviors in youth on the previous seven days.
Minutes of moderate-to-vigorous physical activity out-of-school per week | Change from baseline, to 3 months after the begging if the intervention, end of intervention (after 6-months of baseline assessment), 6 and 12 months follow-up. Specific duration of time over which participant change is assessed: 18 months.
  Youth Activity Profile (YAP): This is a 15 items questionnaire to evaluate psychical activity and sedentary behaviors in youth on the previous seven days.

SECONDARY OUTCOMES:
Eating disturbance | Baseline (before the intervention), 3 months after the begging if the intervention, end of intervention (after 6-months of baseline assessment), 6 and 12 months follow-up. Specific duration of time over which participant is assessed: 18 months.
  Children's Eating Attitudes Test (ChEAT). Higher scores indicate more eating disturbance.
Grazing eating pattern | Baseline (before the intervention), 3 months after the begging if the intervention, end of intervention (after 6-months of baseline assessment), 6 and 12 months follow-up. Specific duration of time over which participant is assessed: 18 months.
  Repetitive Eating Questionnaire (Rep(eat)-Q). Higher scores indicate the existence of a grazing-type eating pattern.
Psychological Distress (depression, anxiety and stress) | Baseline (before the intervention), 3 months after the begging if the intervention, end of intervention (after 6-months of baseline assessment), 6 and 12 months follow-up. Specific duration of time over which participant is assessed: 18 months.
  Depression Anxiety Stress Scales (DASS-21). Higher scores indicating more anxiety, stress and depressive symptomatology.
Health-related quality of life | Baseline (before the intervention), 3 months after the begging if the intervention, end of intervention (after 6-months of baseline assessment), 6 and 12 months follow-up. Specific duration of time over which participant is assessed: 18 months.
  Pediatric Quality of Life Inventory. Higher scores indicate more health-related quality of life.
BMI z-score | Baseline (before the intervention), 3 months after the begging if the intervention, end of intervention (after 6-months of baseline assessment), 6 and 12 months follow-up. Specific duration of time over which participant is assessed: 18 months.
  Calculated by WHO Anthroplus software 3.2.2. version

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Conceição, Ph.D., Principal Investigator — University of Minho, School of Psychology
Locations (2):
- Portugal (2):
  - Centro Hospitalar Universitário do Porto (Centro Materno Infantil do Norte), Porto
  - Centro Hospitalar Universitário de São João, Porto

IPD SHARING:
Plan to Share IPD: No
The type of data to collect include sensitive and personal health information protected by the Portuguese Law.

REFERENCES:
- [Background] Ramalho S, Saint-Maurice PF, Silva D, Mansilha HF, Silva C, Goncalves S, Machado P, Conceicao E. APOLO-Teens, a web-based intervention for treatment-seeking adolescents with overweight or obesity: study protocol and baseline characterization of a Portuguese sample. Eat Weight Disord. 2020 Apr;25(2):453-463. doi: 10.1007/s40519-018-0623-x. Epub 2018 Dec 5. PMID 30519810